CLINICAL TRIAL: NCT03289793
Title: Clinical Evaluation of a Brain Computer Interfaces (BCI)-Based Training of Attention in Children With Attention Deficit Hyperactivity Disorder (ADHD)
Brief Title: NEUROFEEDBACK on Event-Related Potential (ERP)
Acronym: MyB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 69HCL15_0214
Record Dates: First submitted 2017-08-04; First posted 2017-09-21 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: Attention Deficit Disorder with Hyperactivity; ADHD; Children; Inattention; Hyperactivity; Neurofeedback; Neuropsychology
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Spasm

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Children will be assigned to this group in a random fashion according to a ratio 2:1 with respect to group B (see below).
  20 subjects will be included in this group.
  Interventions: Other: Neurofeedback training
- Group B (Active Comparator): Children will be assigned in this group in a random fashion. 10 subjects will be included in this group.
  Interventions: Other: Active Sham control
- Group C (Active Comparator): Will be included in this group children who meet the inclusion criteria and who, with their families, are motivated to participate in the study but cannot claim to be part of groups A or B (because of logistical constraints: living too far away to comply with the frequency of the visits required by the training).
  Group C allows to follow the natural evolution of children with ADHD with no intervention.
  Interventions: Other: Baseline control group

INTERVENTIONS:
Other: Neurofeedback training — Children in group A will receive BCI-based training implemented through original P300-based controlled games.
  They will attend 30 1-hour long training sessions at a pace of 2 sessions per week.
  Each session includes: installation of the child, the EEG system and an eye-tracking system, a 5-minutes relaxation phase, a short EEG recording at rest, a brief reminder of the instructions, 30 minutes of training by playing video games and finally a time for the child to wash her/his hair.
  Moreover, 4 neuropsychological sessions will complement the 30 training sessions. During these sessions neuropsychological tests and quality of life questionnaires will be answered.
  Arms: Group A
Other: Active Sham control — Children in group B will receive a training that is not based on brain activity, but in a blind fashion. They will attend 30 1-hour long training sessions at a pace of 2 sessions per week.
  Each session includes: installation of the child, setting up the EEG and eye-tracking systems, a 5-minutes relaxation phase, short EEG recording at rest, a brief reminder of the instructions, 30 minutes of video game based training and finally a time for the child to wash her/his hair.
  Besides, 4 neuropsychological sessions will complement the 30 training sessions. During these sessions neuropsychological tests and quality of life questionnaires will be performed.
  Arms: Group B
Other: Baseline control group — The children included in this group will not receive any training. They only take part to the 4 neuropsychological sessions. Like others, they will attend 1 neuropsychological session every two months over six months.
  Arms: Group C

SUMMARY:
This project aims to assess the evolution of symptoms in ADHD children from 8 to 17 years, with various types of attention training.

Different groups A, B and C will be evaluated: the first with Neurofeedback training, the second with a similar training but not indexed on brain activity and the third without training.

30 patients will be randomly assigned to groups A and B according to a ratio 2:1.

Others patients who meet the same criteria but for logistical reasons cannot comply with the training constraints will be assigned to group C.

Children included in groups A and B will participate in training sessions (Neurofeedback and control training, respectively) as well as in four evaluation sessions. Children in group C will only participate in evaluation sessions (baseline control group).

Patients of groups A and B will be followed over 6 months: 4 months of training and a follow-up evaluation 2 months after training.

Patients of group C will be followed each 2 months for 6 months. This study uses electro-encephalography measures, serious video game, neuropsychological tests and questionnaires.

It also uses actigraphy measures to evaluate sleep quality.

ELIGIBILITY:
Inclusion Criteria:

* Children and teenagers aged from 8 to 17 years' old
* Children and teenagers with a deficit attention disorder with or without hyperactivity, in the mixed form or in a pure inattentive form according to Diagnostique et Statistique des troubles Mentaux (DSM)-V.
* Children and teenagers having a score in Verbal Comprehension Index (or Index Verbal Reasoning) and Perceptual Reasoning Index (or Index Reasoning fluid) ≥ 80 of WISC IV or V test, not older than two years.
* Children and teenagers without psychostimulant treatment
* Children and teenagers with psychostimulant treatment agreed to achieve a therapeutic break at each visit day and with a stable dose during all the study.
* Children and teenagers whose parents have agreed and signed informed consent form of the study.

Exclusion Criteria:

* Children aged less than 8 and teenagers are more than 18 years' old.
* Children and teenagers having a score in Verbal Comprehension Index (or Index Verbal Reasoning) and Perceptual Reasoning Index (or Index Reasoning fluid) < 80 of WISC IV or V test, not older than two years.
* Children and teenagers with developmental disorder except "Dys" disorders.
* Children and teenagers with pure hyperactivity (without attentional deficit)
* Children and teenagers with epilepsy except benign epilepsies (without brain damage), free of crisis for two years and without treatment.
* Children and teenagers with ADHD with conduct disorders and aggression
* Children and teenagers with ADHD and Tourette's syndrome.
* Patients treated by anti / epilepsy or psychotropic treatments (with the exception of psychostimulant treatment).
* Patients with psychostimulant treatment and whose parents aren't agreed to achieve a therapeutic break at each visit day.
* Patients with visual deficiency uncorrectable with lenses or glasses.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2019-09-09 (Actual); Study Completion 2019-09-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of the relative effect on symptoms of inattention between the two proposed training techniques, A and B, with the ADHD Rating Scale in children with ADHD | every two months over six months.
  Questions with odd numbers interested in the dimension "inattentive" will particularly be studied. The investigator expect an improvement in the type of score: ''ADHD-Inattentive'' children in group A compared to children in Group B. More specifically, he expect to improve responses to questions number 1,3,5,7,9,11,13,15 and 17. By definition, an evolving response would be to move from " 2=Often; 3=Very often" to " 1=Sometimes; 0=Rarely/Never".

SECONDARY OUTCOMES:
Neuropsychological assessments of effects of training on the symptoms of inattention in ADHD children | every months over six months.
  ADHD Rating Scale (questions with odd numbers) will be performed ADHD children from groups A, B and C will be compared
Neuropsychological assessments of effects of training on the symptoms of inattention in ADHD children | every months over six months.
  Bron/Lyon Attention Stability test (BLAST) test will be performed ADHD children from groups A, B and C will be compared
Neuropsychological assessments of effects of training on the symptoms of inattention in ADHD children | every months over six months.
  Wechsler Intelligence Scale for Children (WISC) subtests will be performed ADHD children from groups A, B and C will be compared
Neuropsychological assessments of the effects of the lack of training on the symptoms of inattention in ADHD children | every months over six months.
  Wechsler Intelligence Scale for Children (WISC) will be performed ADHD children from groups A, B and C will be compared
Neuropsychological assessments of the effects of the lack of training on the symptoms of inattention in ADHD children | every months over six months.
  ADHD Rating Scale (questions with odd numbers) will be performed ADHD children from groups A, B and C will be compared
Neuropsychological assessments of the effects of the lack of training on the symptoms of inattention in ADHD children | every months over six months.
  Bron/Lyon Attention Stability test (BLAST) will be performed ADHD children from groups A, B and C will be compared
Compare the effects of the two types of trainings on the hyperactivity symptoms in ADHD children using neuropsychological assessments. | every two months over six months
  ADHD Rating Scale (questions with even numbers), Test d'évaluation de l'Attention (TAP) and Continuous Performance Test (CPT) will be performed ADHD children from groups A, B and C will be compared
neuropsychological assessments of the effects of the two types of trainings on the hyperactivity symptoms in ADHD children | every two months over six months
  ADHD Rating Scale (questions with even numbers) will be performed ADHD children from groups A, B and C will be compared
neuropsychological assessments of the effects of the two types of trainings on the hyperactivity symptoms in ADHD children | every two months over six months
  Test d'évaluation de l'Attention (TAP) will be performed ADHD children from groups A, B and C will be compared
neuropsychological assessments of the effects of the two types of trainings on the hyperactivity symptoms in ADHD children | every two months over six months
  Continuous Performance Test (CPT) will be performed ADHD children from groups A, B and C will be compared
neuropsychological assessments of the effects of the lack of training on the impulsivity symptoms in ADHD children | every two months over six months
  Continuous Performance Test (CPT) will be performed ADHD children from groups A, B and C will be compared
neuropsychological assessments of the effects of the lack of training on the impulsivity symptoms in ADHD children | every two months over six months
  Test d'évaluation de l'Attention (TAP) will be performed ADHD children from groups A, B and C will be compared
neuropsychological assessments of the effects of the lack of training on the impulsivity symptoms in ADHD children | every two months over six months
  ADHD Rating Scale (questions with even numbers) will be performed ADHD children from groups A, B and C will be compared
neuropsychological assessments of the effects of the lack of training on the hyperactivity symptoms in ADHD children | every two months over six months
  Continuous Performance Test (CPT) will be performed ADHD children from groups A, B and C will be compared
neuropsychological assessments of the effects of the lack of training on the hyperactivity symptoms in ADHD children | every two months over six months
  ADHD Rating Scale (questions with even numbers) will be performed ADHD children from groups A, B and C will be compared
neuropsychological assessments of the effects of the lack of training on the hyperactivity symptoms in ADHD children | every two months over six months
  Test d'évaluation de l'Attention (TAP) will be performed ADHD children from groups A, B and C will be compared
Quantify whether the changes in inattentive symptoms in groups A (Neurofeedback training) correlate with changes in specific EEG parameter, namely the P300 wave. | every two months over six months
  ADHD Rating Scale (questions with odd numbers) will be evaluated ADHD children of groups A, B and C will be compared
Quantify whether the changes in inattentive symptoms in groups A (Neurofeedback training) correlate with changes in specific EEG parameter, namely the P300 wave. | every two months over six months
  TAP will be evaluated ADHD children of groups A, B and C will be compared
Quantify whether the changes in inattentive symptoms in groups A (Neurofeedback training) correlate with changes in specific EEG parameter, namely the P300 wave. | every two months over six months
  CPT will be evaluated ADHD children of groups A, B and C will be compared
Quantify whether the changes in inattentive symptoms in groups A (Neurofeedback training) correlate with changes in specific EEG parameter, namely the P300 wave. | every two months over six months
  BLAST will be evaluated ADHD children of groups A, B and C will be compared
Quantify whether the changes in inattentive symptoms in groups A (Neurofeedback training) correlate with changes in specific EEG parameter, namely the P300 wave. | every two months over six months
  Attention and Distractibility Questionnaire (for children) will be evaluated ADHD children of groups A, B and C will be compared
Quantify whether the changes in inattentive symptoms in groups B (Neurofeedback training) correlate with changes in specific EEG parameter, namely the P300 wave. | every two months over six months
  ADHD Rating Scale (questions with odd numbers)will be evaluated ADHD children of groups A, B and C will be compared
Quantify whether the changes in inattentive symptoms in groups B (Neurofeedback training) correlate with changes in specific EEG parameter, namely the P300 wave. | every two months over six months
  TAP will be evaluated ADHD children of groups A, B and C will be compared
Quantify whether the changes in inattentive symptoms in groups B (Neurofeedback training) correlate with changes in specific EEG parameter, namely the P300 wave. | every two months over six months
  CPT will be evaluated ADHD children of groups A, B and C will be compared
Quantify whether the changes in inattentive symptoms in groups B (Neurofeedback training) correlate with changes in specific EEG parameter, namely the P300 wave. | every two months over six months
  BLAST will be evaluated ADHD children of groups A, B and C will be compared
Quantify whether the changes in inattentive symptoms in groups B (Neurofeedback training) correlate with changes in specific EEG parameter, namely the P300 wave. | every two months over six months
  Attention and Distractibility Questionnaire (for children) will be evaluated ADHD children of groups A, B and C will be compared
Quantify whether the changes in inattentive symptoms in groups C (Neurofeedback training) correlate with changes in specific EEG parameter, namely the P300 wave. | every two months over six months
  ADHD Rating Scale (questions with odd numbers) will be evaluated ADHD children of groups A, B and C will be compared
Quantify whether the changes in inattentive symptoms in groups C (Neurofeedback training) correlate with changes in specific EEG parameter, namely the P300 wave. | every two months over six months
  TAP will be evaluated ADHD children of groups A, B and C will be compared
Quantify whether the changes in inattentive symptoms in groups C (Neurofeedback training) correlate with changes in specific EEG parameter, namely the P300 wave. | every two months over six months
  CPT will be evaluated ADHD children of groups A, B and C will be compared
Quantify whether the changes in inattentive symptoms in groups C (Neurofeedback training) correlate with changes in specific EEG parameter, namely the P300 wave. | every two months over six months
  BLAST will be evaluated ADHD children of groups A, B and C will be compared
Quantify whether the changes in inattentive symptoms in groups C (Neurofeedback training) correlate with changes in specific EEG parameter, namely the P300 wave. | every two months over six months
  Attention and Distractibility Questionnaire (for children) will be evaluated ADHD children of groups A, B and C will be compared
Quantify the evolution of the classical Neurofeedback biomarkers Slow Cortical Potential (SCP)) | every two months over six months
  ADHD Rating Scale (questions with odd numbers) will be evaluated ADHD children of groups A, B and C will be compared
Quantify the evolution of the classical Neurofeedback biomarkers Slow Cortical Potential (SCP)) | every two months over six months
  TAP will be evaluated ADHD children of groups A, B and C will be compared
Quantify the evolution of the classical Neurofeedback biomarkers Slow Cortical Potential (SCP)) | every two months over six months
  BLAST will be evaluated ADHD children of groups A, B and C will be compared
Quantify the evolution of the classical Neurofeedback biomarkers Slow Cortical Potential (SCP)) | every two months over six months
  Attention and Distractibility Questionnaire (child) will be evaluated ADHD children of groups A, B and C will be compared
Assess whether the classical Neurofeedback biomarkers correlate with the evolution of behavioral and primary neurophysiological measures (P300) in all groups. | every two months over six months
  ADHD Rating Scale (questions with odd numbers) will be evaluated ADHD children of groups A, B and C will be compared
Assess whether the classical Neurofeedback biomarkers correlate with the evolution of behavioral and primary neurophysiological measures (P300) in all groups. | every two months over six months
  TAP will be evaluated ADHD children of groups A, B and C will be compared
Assess whether the classical Neurofeedback biomarkers correlate with the evolution of behavioral and primary neurophysiological measures (P300) in all groups. | every two months over six months
  BLAST will be evaluated ADHD children of groups A, B and C will be compared
Assess whether the classical Neurofeedback biomarkers correlate with the evolution of behavioral and primary neurophysiological measures (P300) in all groups. | every two months over six months
  Attention and Distractibility Questionnaire (child) will be evaluated ADHD children of groups A, B and C will be compared
Quantify the evolution of the classical Neurofeedback biomarkers Theta/Beta Ratio (TBR) | every two months over six months
  ADHD Rating Scale (questions with odd numbers) will be evaluated ADHD children of groups A, B and C will be compared
Quantify the evolution of the classical Neurofeedback biomarkers Theta/Beta Ratio (TBR) | every two months over six months
  TAP will be evaluated ADHD children of groups A, B and C will be compared
Quantify the evolution of the classical Neurofeedback biomarkers Theta/Beta Ratio (TBR) | every two months over six months
  BLAST will be evaluated ADHD children of groups A, B and C will be compared
Quantify the evolution of the classical Neurofeedback biomarkers Theta/Beta Ratio (TBR) | every two months over six months
  Attention and Distractibility Questionnaire (child) will be evaluated ADHD children of groups A, B and C will be compared
Assess whether the classical Neurofeedback biomarkers TBR correlate with the evolution of behavioral and primary neurophysiological measures (P300) in all groups. | every two months over six months
  ADHD Rating Scale (questions with odd numbers) will be evaluated ADHD children of groups A, B and C will be compared
Assess whether the classical Neurofeedback biomarkers TBR correlate with the evolution of behavioral and primary neurophysiological measures (P300) in all groups. | every two months over six months
  TAP will be evaluated ADHD children of groups A, B and C will be compared
Assess whether the classical Neurofeedback biomarkers TBR correlate with the evolution of behavioral and primary neurophysiological measures (P300) in all groups. | every two months over six months
  BLAST will be evaluated ADHD children of groups A, B and C will be compared
Assess whether the classical Neurofeedback biomarkers TBR correlate with the evolution of behavioral and primary neurophysiological measures (P300) in all groups. | every two months over six months
  Attention and Distractibility Questionnaire (child) will be evaluated ADHD children of groups A, B and C will be compared
Quantify the evolution of the classical Neurofeedback biomarkers Sensori-Moteur Rythm (SMR) | every two months over six months
  ADHD Rating Scale (questions with odd numbers) will be evaluated ADHD children of groups A, B and C will be compared
Quantify the evolution of the classical Neurofeedback biomarkers Sensori-Moteur Rythm (SMR) | every two months over six months
  TAP will be evaluated ADHD children of groups A, B and C will be compared
Quantify the evolution of the classical Neurofeedback biomarkers Sensori-Moteur Rythm (SMR) | every two months over six months
  BLAST will be evaluated ADHD children of groups A, B and C will be compared
Quantify the evolution of the classical Neurofeedback biomarkers Sensori-Moteur Rythm (SMR) | every two months over six months
  Attention and Distractibility Questionnaire (child) will be evaluated ADHD children of groups A, B and C will be compared
Assess whether the Neurofeedback biomarkers SMR correlate with the evolution of behavioral and primary neurophysiological measures (P300) in all groups. | every two months over six months
  ADHD Rating Scale (questions with odd numbers)will be evaluated ADHD children of groups A, B and C will be compared
Assess whether the Neurofeedback biomarkers SMR correlate with the evolution of behavioral and primary neurophysiological measures (P300) in all groups. | every two months over six months
  TAP will be evaluated ADHD children of groups A, B and C will be compared
Assess whether the Neurofeedback biomarkers SMR correlate with the evolution of behavioral and primary neurophysiological measures (P300) in all groups. | every two months over six months
  BLAST will be evaluated ADHD children of groups A, B and C will be compared
Assess whether the Neurofeedback biomarkers SMR correlate with the evolution of behavioral and primary neurophysiological measures (P300) in all groups. | every two months over six months
  Attention and Distractibility Questionnaire (child) will be evaluated ADHD children of groups A, B and C will be compared
Evaluate the impact of the trainings on the sleep quality in ADHD children. | every two months over six months.
  Sleep questionnaires will be distributed ADHD children in groups A, B and C will be compared.
Evaluate the impact of the trainings on the sleep quality in ADHD children. | every two months over six months.
  The sleep data may also be collected using an actigraph (ancillary study). ADHD children in groups A, B and C will be compared.
Evaluating the impact of the trainings on the quality of life in ADHD children. | every two months over six months
  The Child Behavior CheckList (CBCL) questionnaire will be performed
  Groups A, B and C will be compared.
Evaluating the impact of the trainings on the quality of life in ADHD children. | every two months over six months
  Information about the quality of life will be also collected in a logbook by family members and provided at each visit.
  Groups A, B and C will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Alexis ARZIMANOGLOU, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Bron, France